CLINICAL TRIAL: NCT03308487
Title: Evaluation and Comparison of the Efficacy of 1000 and 2000 IU/d Vitamin D Supplementation During Pregnancy on Maternal and Newborn Vitamin D Status and Pregnancy Outcomes
Brief Title: Vitamin D Supplementation and Pregnancy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tirang R. Neyestani, Ph.D. (Other)
Collaborators: National Nutrition and Food Technology Institute (Other)
Responsible Party: Sponsor-Investigator, Tirang R. Neyestani, Ph.D., Professor (research), National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IR.SBMU.RETECH.1395.631
Record Dates: First submitted 2017-01-13; First posted 2017-10-12 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Maternal Vitamin D Status
Keywords: Vitamin D; pregnancy
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3 (1000 IU) (Active Comparator): group 1
  Interventions: Dietary Supplement: vitamin D3 (1000 IU)
- vitamin D3 (2000 IU) (Active Comparator): group 2
  Interventions: Dietary Supplement: Vitamin D3 (2000 IU)

INTERVENTIONS:
Dietary Supplement: vitamin D3 (1000 IU)
  Arms: vitamin D3 (1000 IU)
Dietary Supplement: Vitamin D3 (2000 IU)
  Arms: vitamin D3 (2000 IU)

SUMMARY:
Groups (group 1 receives 1000 IU vitamin D and group 2 receives 2000 IU vitamin D) through a random allocation. It is necessary to mention that all cases in each group could be able to receive the current supplementation during pregnancy (Folic acid, iron and multivitamin and calcium). This study aimed to evaluate the efficacy of two doses of vitamin D supplementation (1000 and 2000 IU/d) during pregnancy on maternal and newborn vitamin D status and metabolic profile including lipid profile (serum concentration of total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), triglyceride(TG)), glucose homeostasis (fasting glucose, insulin, insulin resistance (HOMA-IR)) and inflammatory and oxidative stress (OS) markers and pregnancy outcomes including gestational diabetes, preeclampsia, preterm delivery, abortion, cesarian section, and also anthropometric data and apgar score of infants compared with placebo.

DETAILED DESCRIPTION:
In this randomized controlled trial, 84 pregnant women aged at 18-40 years with gestational age of <12 weeks will be recruited and divided into 2 groups.

Demographic, socioeconomic and lifestyle data as well as blood samples and urine samples will be collected at baseline and in the last month of pregnancy. Moreover the cord blood will be collected at birth.

Fasting blood glucose, insulin resistance (HOMA-IR), insulin, lipid profile (serum concentration of total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), triglyceride(TG)), inflammatory (IL-1β, IL-6, TNF-α, hs-CRP) and oxidative stress markers (MDA, TAC), calcium:creatinine ratio are going to be evaluated at the beginning and in the end of the interventional period in pregnant women. Inflammatory (IL-1β, IL-6, Tumor Necrosis Factor (TNF-α), hs-CRP) and oxidative stress markers (MDA, TAC) will be determined in cord blood as well.

ELIGIBILITY:
Inclusion Criteria:

* maternal age of 18-40 years,
* gestational age of 12 weeks or less,
* singleton pregnancies,
* mothers supposed to have normal pregnancy and not having preexisting diseases like hypertension, or cardiac, renal, hepatic, autoimmune , rheumatoid arthritis and digestive disease, or endocrinological disorders including diabetes (type 1 or type 2 diabetes), parathyroid disorders, and thyroid disorder,
* not receiving dietary supplements including vitamin D (>600 IU/d), or omega-3 within the past 3 months before the intervention,
* not taking medications that could potentially influence vitamin D metabolism,
* willingness to participate in the study.

Exclusion Criteria:

* Participants who do not meet the inclusion criteria,
* those who diagnosed to have fasting blood sugar (FBS)>92 at first blood sampling and/or blood pressure > 140/90 mmHg at the first visit,
* using extra vitamin D3 supplement and/or omega-3 and/or other medications that could potentially influence vitamin D metabolism,
* fetal anomaly,
* poor adherence to the study protocol,
* unwillingness to continue the intervention.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The changes in maternal vitamin D status from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of 25(OH) D will be measured during the first trimester and last month of pregnancy.

SECONDARY OUTCOMES:
The changes in serum concentration of fasting blood glucose from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of fasting blood glucose will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of insulin from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of insulin will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of total cholesterol (TC) from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of total cholesterol (TC) will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of low-density lipoprotein cholesterol (LDL-C) from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of low-density lipoprotein cholesterol (LDL-C) will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of high-density lipoprotein cholesterol (HDL-C) from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of high-density lipoprotein cholesterol (HDL-C) will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of triglyceride(TG) from first trimester to last month of pregnancy | baseline and 6-8 months
  The serum concentration of triglyceride(TG) will be measured during the first trimester and last month of pregnancy.
The changes in systolic blood pressure from first trimester to last month of pregnancy | baseline and 6-8 months
  systolic and diastolic blood pressure will be measured by a training physician
The changes in diastolic blood pressure from first trimester to last month of pregnancy | baseline and 6-8 months
  systolic and diastolic blood pressure will be measured by a training physician
preeclampsia | 2-5 months
  Preeclampsia characterized by high blood pressure begins after 20 weeks of pregnancy in women whose blood pressure had been normal.
Preterm delivery | 5-8 months
  A premature birth is a birth that takes place before the start of the 37th week of pregnancy.
Spontaneous abortion | 2-5 months
  Spontaneous abortion is the natural death of an embryo or fetus before 20 weeks of gestation.
The changes in cellular secretion of interleukin 1 from first trimester to last month of pregnancy | baseline and 6-8 months
  The status of interleukin 1 will be measured during the first trimester and last month of pregnancy.
The changes in cellular secretion of interleukin 6 from first trimester to last month of pregnancy | baseline and 6-8 months
  The status of interleukin 6 will be measured during the first trimester and last month of pregnancy.
The changes in cellular secretion of interleukin 10 from first trimester to last month of pregnancy | baseline and 6-8 months
  The status of interleukin 10 will be measured during the first trimester and last month of pregnancy.
The changes in cellular secretion of TNF-a from first trimester to last month of pregnancy | baseline and 6-8 months
  The status of TNF-a will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of hs-CRP from first trimester to last month of pregnancy | baseline and 6-8 months
  The status of hs-CRP will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of MDA (Malondialdehyde) from first trimester to last month of pregnancy | baseline and 6-8 months
  the serum concentration of MDA (Malondialdehyde) will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of TAC from first trimester to last month of pregnancy | baseline and 6-8 months
  the serum concentration of TAC will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of parathyroid hormone (PTH) from first trimester to last month of pregnancy | baseline and 6-8 months
  the serum concentration of parathyroid hormone (PTH) will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of calcium from first trimester to last month of pregnancy | baseline and 6-8 months
  the serum concentration of calcium will be measured during the first trimester and last month of pregnancy.
The changes in serum concentration of phosphate from first trimester to last month of pregnancy | baseline and 6-8 months
  the serum concentration of phosphate will be measured during the first trimester and last month of pregnancy.
Apgar score | 6-8 months
  The Apgar score is a quick evaluation of one minute and five minutes after birth which tests the birthing process and readiness of newborn to meet the world without additional medical assistance.
The weight measures of newborn | 6-8 months
  The data of anthropometric measures including weight will be measured.
The height measures of newborn | 6-8 months
  The data of anthropometric measures including height will be measured.
The head circumference measures of newborn | 6-8 months
  The data of anthropometric measures including head circumference will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R Neyestani, PhD, Study Chair — National Nutrition and Food Technology Research Institute
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Motamed S, Nikooyeh B, Kashanian M, Chamani M, Hollis BW, Neyestani TR. Evaluation of the efficacy of two doses of vitamin D supplementation on glycemic, lipidemic and oxidative stress biomarkers during pregnancy: a randomized clinical trial. BMC Pregnancy Childbirth. 2020 Oct 14;20(1):619. doi: 10.1186/s12884-020-03311-1. PMID 33054794